CLINICAL TRIAL: NCT05262166
Title: Opioid-Free Anaesthesia During Prolonged Orthotopic Urinary Bladder Diversion Surgery: A Prospective Randomized Comparative Study.
Brief Title: Opioid Free Anesthesia in Prolonged Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS.21.10.1699(date 21/11/2021)
Record Dates: First submitted 2022-02-04; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Cancer, Bladder
Keywords: Opioid-Free Anaesthesia; Prolonged Orthotopic Urinary Bladder Diversion Surgery; Intrathecal dexmedetomidine
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural Fentanyl group: (No Intervention): Epidural Fentanyl group: using an epidural catheter technique with epidural catheter set, and at L1-2 insertion level directed up to cover up to T6 sensory level, 5ml of bupivacaine 0.5%plus 50 micrograms fentanyl in a total volume of 40 ml added saline 0.9% (epidural injection of bolus of total Volume of 15 ml of 0.0625%bupivacaine with 1.25Mcg/ml fentanyl) then for next G anaesthesia hours to run in a 3-5 ml/h epidural infusion rate.
- Intrathecal dexmedetomidine group: (Experimental): Intrathecal dexmedetomidine plus heavy bupivacaine then general A
  Interventions: Drug: INTRATHECAL dexmedetomidine INJECTION

INTERVENTIONS:
Drug: INTRATHECAL dexmedetomidine INJECTION — intrathecal bolus of 3ml bupivacaine 0.5% (15mg) plus 10 micrograms dexmedetomidine at 2-3 or 3-4 spinal level.
  Arms: Intrathecal dexmedetomidine group:

SUMMARY:
this study is designed to compare intrathecal bolus of bupivacaine-dexmedetomidine versus continuous epidural fentanyl infusion in providing effective operative analgesia, intraoperative hemodynamic stability and less postoperative cumulative opioid induced complications in orthotopic urinary bladder diversion prolonged surgery.

The hypothesis Intrathecal bolus of bupivacaine-dexmedetomidine could replace continuous epidural fentanyl infusion and would be an enough intraoperative analgesic modality with good intraoperative hemodynamic stability and less postoperative complications in orthotopic urinary bladder diversion patients.

Aim of the work The aim of this protocol is to document that intrathecal bolus of bupivacaine-dexmedetomidine analgesia (a low coast analgesic modality) can replace continuous epidural fentanyl infusion analgesic modality with effective operative analgesia, intraoperative hemodynamic stability and less postoperative cumulative opioid induced complications in orthotopic urinary bladder diversion prolonged surgery.

DETAILED DESCRIPTION:
Opioid-free anaesthesia is becoming a popular technique among clinicians. The technique involves administering anaesthesia without any intraoperative systemic, neuraxial or intracavitary opioid It helps in avoiding the opioids during the perioperative period. Opioid-free anaesthesia can be performed along with loco-regional analgesia for better pain control, though it is not always mandatory Spinal bupivacaine-dexmedetomidine can produce intraoperative prolonged continuous analgesia in abdominal surgeries. On the other hand, the stability of continuous epidural fentanyl infusion would produce hemodynamic stability with effective analgesia in orthotopic urinary bladder diversion as an analgesia technique during prolonged abdominal surgery free of nephrotoxic drugs such as NSAIDs. Lipophilic opioids such as fentanyl remain longer within the epidural space by partitioning into epidural fat and thus are found in lower concentrations in cerebrospinal fluid compared with hydrophilic opioids such as morphine. During prolonged infusion of lipophilic opioids such as fentanyl and sufentanyl, the plasma concentration and analgesic effect of these drugs are similar to that of an intravenous infusion .

Titration of epidural local anesthetic and opioid concentrations must be performed to attain a balance between providing optimal analgesia and avoiding hemodynamic instability. The addition of fentanyl does not prolong the sensory and motor block characteristics of dexmedetomidine .

Intrathecal dexmedetomidine is superior to intrathecal magnesium sulfate (MgSO4) during caesarean section with regard to duration of analgesia, pain severity and stress hormone levels. Dexmedetomidine has a rapid onset and longer duration of sensory block compared to MgSO4 .

Paramasivan and his colleagues documented that intrathecal dexmedetomidine has prolonged postoperative analgesic duration, reduced 24 hours pain intensity and reduced the incidence of shivering without an increase in other adverse effects compared to placebo .

Using dexmedetomidine as an adjuvant to bupivacaine for spinal anesthesia in lower limb surgeries has longer duration of sensory and motor block and longer postoperative analgesia .

Mazy and his colleagues documented that intrathecal dexmedetomidine 10 micrograms (mic) and bupivacaine 20 milligram with or without fentanyl 25 mic were suitable for long orthopedic procedures within 6 hours duration. The addition of fentanyl does not prolong the sensory and motor block characteristics of dexmedetomidine. In favor of dexmedetomidine-fentanyl combination was the less hypotension and less sedative requirement .

Epidural fentanyl administered by a continuous infusion can provide an efficient postoperative analgesia and is responsible for a moderate ventilatory depression .

Patel Nagar and his colleagues documented that intrathecal dexmedetomidine of 10 micrograms when compared to lower doses as an adjuvant to hyperbaric bupivacaine significantly prolongs the duration of sensory block, motor block, and analgesia. A disproportionate increase in the duration of analgesia and motor block produces both clinically and statistically significant prolongation of the duration of differential analgesia. Addition of 10 micrograms of intrathecal dexmedetomidine is associated with fewer requirements of postoperative analgesics in patients undergoing lower abdominal and lower limb surgeries without any significant increase in the incidence of side effects .

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for orthotopic urinary bladder diversion prolonged surgery procedures.
2. American society of Anaethesiologists (ASA I-II).
3. Both sexes.
4. Age 18 - 70 years.

Exclusion Criteria:

1. Patient refusal.
2. Hypersensitivity to amide local anesthetics or opioids as fentanyl.
3. General contraindications to spinal and epidural anaesthesia as thrombocytopenia, coagulopathy and severe dehydration.
4. Uncompensated Cardiac or hepatic patients.
5. Renal failure or respiratory failure patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2022-08-10 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Total postoperative ANALGESIC fentanyl DOSE | first 24 hours in both groups.
  Total postoperative intravenous fentanyl requirements in the first twinty four hours after spinal dexmedetomedine

CONTACTS AND LOCATIONS:
Overall Officials: MOHAMED GHANEM, professor, Study Director — Urology Nephrology center, Faculty of Medicine, Mansoura Univeristy
Locations (1):
- Medicine, Al Mansurah, Dakahlia Governorate, Egypt